CLINICAL TRIAL: NCT04090515
Title: Project Health Intervention Among Latinx Adults in Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Michael J. Zvolensky, Ph.D., Principal Investigator, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00001757
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Obesity
Keywords: Obesity; Eating; Physical Activity; Exercise
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: If participant meets eligibility criteria, the participant will be block randomized to one of two conditions: either (1) active (n = 12) or (2) educational video control (n = 6)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project Health (Experimental): Project Health has three aims: 1) encourage participants to explore the costs of obesity, an unhealthy diet, and sedentary behavior and the benefits of physical fitness, a healthy diet, and regular exercise; 2) help participants gradually reduce caloric intake and increase physical activity, such that the participant reaches energy balance (i.e., is not eating more calories than they need); and 3) reduce attitudinal and behavioral risk factors for eating disorders and obesity. The intervention will be administered in Spanish.
  Interventions: Behavioral: Project Health
- Educational Video Control (Placebo Comparator): The educational video control condition will include an educational video series on obesity in Spanish.
  Interventions: Other: Educational Video Control

INTERVENTIONS:
Behavioral: Project Health — This intervention involves a one-hour group meeting for six consecutive weeks.
  Arms: Project Health
Other: Educational Video Control — This intervention involves a one-hour educational video control viewing for six consecutive weeks.
  Arms: Educational Video Control

SUMMARY:
The proposed study will examine acceptability/feasibility and establish initial estimates of effect sizes of an existing intervention (Project Health) on a sample of young adult Latinx individuals in a primary health care setting. Project Health intervention involves making small, participant-identified, gradually increasing improvements to their dietary intake and exercise.

DETAILED DESCRIPTION:
The primary goal of the research study is to investigate the acceptability/feasibility and establish initial estimates of effect sizes of Project Health that addresses dietary intake and exercise to reduce BMI, eating disorder symptoms, negative affect, and food cravings at post-intervention. To address this aim, the research will involve a randomized control trial that will employ a longitudinal experimental design that will involve: (a) phone-screener (pre-screener); (b) baseline appointment consisting of a pre-intervention assessment (eligibility); (c) 6-week intervention (randomized to Project Health or Video Control); (d) 3-month follow-up, (e) 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported Hispanic/Latino ethnicity
* Ability to read, write, and communicate in Spanish
* Report concern about their weight
* Affirming weight gain within the past year and/or belief that there is room for improvement in diet/exercise habits.

Exclusion Criteria:

* Limited mental competency
* Inability to provide, voluntary, written consent
* Endorsement of current or past psychotic-spectrum symptoms
* A reported BMI of < 20 or > 30
* Current diagnosis of anorexia nervosa, bulimia nervosa, or binge eating disorder
* Active suicidality.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index | Assess change from baseline to 3-month follow-up and 1-year follow-up.
  Body mass index will be used to assess obesity. For the current study objective height and weight measurements will be obtained from each participant. BMI will be calculated per World Health Organization (WHO) recommendations based on measured weight and height ([weight (pounds)]/[height (inches)2 x 703]) with lower values indicating better outcomes.

SECONDARY OUTCOMES:
Eating Disorder Diagnostic Scale | Assess change from baseline to 3-month follow-up and 1-year follow-up.
  The Eating Disorder Diagnostic Interview is a 23-item questionnaire used to assess assesses symptoms of anorexia nervosa, bulimia nervosa, and binge eating disorder, which will allow us to exclude participants with these disorders. It also provides a continuous measure of overall eating disorder symptoms.
Positive and Negative Affect Schedule | Assess change from baseline to 3-month follow-up and 1-year follow-up.
  The Positive and Negative Affect Schedule will assess the extent that participants experience 20 different feelings and emotions (e.g., distressed, excited) on a 5-point Likert-type scale ranging from 1 (very slightly or not at all) to 5 (extremely). The PANAS subscale negative affectivity will be summed (possible range = 41 - 205) and lower scores indicating better outcomes.
Food Craving Inventory | Assess change from baseline to 3-month follow-up and 1-year follow-up.
  The Food Craving Inventory is a 28-item self-report instrument that is widely used to measure overall food cravings as well as craving for sweet food, high-fat food, starchy food, and fast-food (FCI-FF). Items are rated on a scale from 1 (Never) to 5 (Always/Almost every day) and averaged with lower scores indicating better outcomes (possible range = 1-5).

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Zvolensky, Ph.D., Principal Investigator — University of Houston
Locations (1):
- RESTORE Laboratory: Research on Emotion, Substance Treatment Outcomes, and Racial Equity, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No